CLINICAL TRIAL: NCT00919009
Title: A Phase II Study of the Combination of TACE and Sorafenib for Patients With Unresectable Hepatocellular Carcinoma in National Cancer Center Korea (COTSUN Korea Trial)
Brief Title: Combination of Transcatheter Arterial Chemoembolization (TACE) and Sorafenib for Patients With Unresectable Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Joong-Won Park, Chief of Hepato - Biliary - Pancreatic Cancer Branch, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: COTSUN Korea Trial
Record Dates: First submitted 2009-04-27; First posted 2009-06-11 (Estimated); Last update posted 2012-05-30 (Estimated); Status verified 2009-06

CONDITIONS: Carcinoma, Hepatocellular
Keywords: TACE; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafeinb (Experimental): Oral sorafenib (400 mg BID) will be start the 3 day after the first TACE treatment and will continue until the patient shows disease progression, until unacceptable toxicity occurs, or until study termination.
  Interventions: Procedure: TACE (Transcatheter Arterial Chemoembolization )

INTERVENTIONS:
Procedure: TACE (Transcatheter Arterial Chemoembolization ) — TACE will be performed according to National Cancer Center protocol:
  Briefly, an arterial catheter was inserted into the femoral artery by the Seldinger method and placed in the hepatic artery. Tumor feeding vessels were superselected where possible, the catheter was inserted to the level of the segmental arteries, subsegmental arteries, or lobar branches, and a solution containing 20-60 mg of doxorubicin hydrochloride (ADM; Dong-a Pharmacy, Seoul, Korea) and 2-20 mLof iodized oil (lipiodol) was infused through the catheter (5 French) or microcatheter (2.8 or 3 French). The dosage of doxorubicin and lipiodol was determined according to the tumor size, the presence of arteriovenous shunts or extrahepatic collateral vessels, and the underlying liver functions

SUMMARY:
Most HCC patients are diagnosed at advanced stages in Korea, transcatheter arterial chemoembolization is considered a key modality for palliative treatment in these HCC patients. TACE is currently one of the mainstays of palliative treatments worldwide for patients with inoperable HCC and it has shown survival benefits in patients with unresectable HCC. TACE consists primarily of directly targeted chemotherapy and embolization of arteries feeding the tumors, inevitably resulting in a hypoxic insult to HCC and surrounding liver tissues. Ischemic injury after TACE has been found to induce the upregulation of circulating vascular endothelial growth factor (VEGF), which is essential for tumor growth, invasion and metastasis in patients with HCC. Recent studies have shown a significant correlation between pre-TACE level of circulating VEGF or VEGF upregulation after TACE and HCC characteristics, including tumor size, vascular invasion, and metastasis. TACE consists primarily of directly targeted chemotherapy and embolization of arteries feeding the tumors, inevitably resulting in a hypoxic insult to HCC and surrounding liver tissues. Central tumor hypoxia was found to upregulate proangiogenic growth factors, which are potent mediators of tumor angiogenesis. Therefore, expression of circulating or tissue VEGF was enhanced after TACE in patients or animals with HCC, and there could be some probability of adverse effects of TACE in HCC patients.

In addition, the investigators demonstrated that a transient increment of serum VEGF level after TACE was significantly correlated with poor outcomes of tumor progression, especially outcomes relevant to distant metastasis.

Therefore, these findings suggest a rationale for applying adjuvant therapy with anti-angiogenesis agent additional treatment of anti-angiogenesis after TACE or during TACE in a selected group of patients HCC.

The aim of this study is to evaluate efficacy and safety of sorafenib 400 mg bid with TACE in patients with unresectable and/or inoperable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide signed written informed consent
* Patients with clinical or histological diagnosis of HCC based on the guidelines of the Korean Liver Cancer Study Group and the National Cancer Center Korea
* Patients with at least one, bi-dimensionally measurable lesion by multiphasic spiral CT scan or dynamic contrast-enhanced MRI
* Patients with stage III or IVa HCC according to modified International Union Against Cancer TNM staging criteria without invasion in main portal vein, or inferior vena cava and extrahepatic metastasis and size of largest tumor 10cm at study entry
* Patients with unresectable or inoperable HCC indicated for TACE as a treatment of choice according to the guidelines of the Korean Liver Cancer Study Group and the National Cancer Center Korea
* Age ≥ 20 years
* ECOG Performance Status of 0 or1
* Child-Pugh class A or B (Child-Pugh score 7)
* Life expectancy of at least 16 weeks
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 7 days prior to screening:

  * Hb ≧ 9g/dl
  * Absolute neutrophil count > 1000/mm3
  * Platelet count ≧ 60x109/L
  * Adequate clotting function: INR < 1.5
  * Hepatic: AST or ALT < 5 X ULN
  * Renal: serum creatinine < 1.5 x ULN
  * Bilirubin ≦ 3mg/dL

Exclusion Criteria:

* Patients with diffuse infiltrative type of HCC that are poorly defined
* Presence of hepatic encephalopathy and intractable ascites
* Active clinically serious infections (> grade 2 NCI-CTC version 3.0), including spontaneous bacterial peritonitis
* History of esophageal or gastric variceal bleeding
* Patients who are on a liver transplant list
* History of cardiac disease: congestive heart failure > NYHA class 2; active coronary artery disease (myocardial infarction more than 6 months prior to study entry is allowed), cardiac arrythmias requiring anti-arrythmic therapy or uncontrolled hypertension and diabetes mellitis
* History of AIDS/HIV infection -Patients with seizure disorder requiring medication (such as steroids or anti- epileptics)
* History of organ allograft
* Patients with evidence or history of bleeding diathesis
* Patients undergoing renal dialysis
* Previous or concurrent cancer that is distinct in primary site or histology from the cancer being evaluated in this study except cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1) or any cancer curatively treated > 3 years prior to study entry.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1Year
Time to progression (TTP) in patients treated with TACE plus sorafenib | 1year

SECONDARY OUTCOMES:
Progression free survival (PFS) will be evaluated | 1year
Overall response rate will be evaluated | 1year

CONTACTS AND LOCATIONS:
Overall Officials: Joong-Won Park, Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Seoul, South Korea